CLINICAL TRIAL: NCT07242222
Title: Evaluating the Safety and Efficacy of Erdosteine in the Treatment of Nonalcoholic Fatty Liver Disease Patients
Brief Title: Erdosteine in the Treatment of Nonalcoholic Fatty Liver Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98467
Record Dates: First submitted 2025-11-15; First posted 2025-11-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver | interventions — Standard of Care; erdosteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 25 patients received the standard conventional therapy in addition to placebo for 3 months.
  Interventions: Other: Standard Therapy
- Erdosteine group (Active Comparator): 25 patients were given the standard conventional therapy plus erdostiene 300 mg two times daily.
  Interventions: Other: Standard Therapy; Drug: Erdosteine

INTERVENTIONS:
Other: Standard Therapy — • The standard conventional therapy in both groups included regular exercise in the form of any physical activity as walking, cycling, etc. for 30-45 minutes minimum 5 days per week in addition to calorie restriction in overweight and obese patients (1200-1500 and 1000-1200 kcal/day for men and women, respectively).
Drug: Erdosteine — Erdosteine is an oral mucoactive agent with antioxidant and anti-inflammatory properties that also reduces bacterial adhesiveness and enhances the effects of antibiotic therapy, all of these properties may be useful for the prevention and treatment of COPD exacerbations
  Arms: Erdosteine group

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a global public health concern, and the leading cause of chronic liver disease, especially in developed countries (1). NAFLD is characterized by lipid accumulation in the liver not attributed to other causes. NAFLD is characterized by excessive hepatic fat accumulation without other recognized causes of increased fat content (e.g., alcohol, virus, drugs, and autoimmunity). According to the Clinical Practice Guidelines of the European Association for the Study of the Liver, the diagnosis of NAFLD requires the exclusion of daily alcohol consumption >30 g for men and >20 g for women

ELIGIBILITY:
Inclusion Criteria:

Either male or female adult patients (>18 years) with fatty liver diagnosis by using upper abdominal ultrasound echography (US).

Exclusion Criteria:

Pregnant and/or lactating women, excessive alcohol use (defined as an average alcohol intake > 30 g per day in men and > 20 g per day in women).

Other etiology of chronic liver diseases such as viral hepatitis, drug-induced hepatitis, and autoimmune hepatitis.

Patients suffering from chronic kidney disease, hyper/hypoparathyroidism. Hypersensitivity to erdostiene.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
The change in the degree of steatosis in the ultrasound (US) is the primary endpoint. | 3 months
  The change in the degree of steatosis in the US is the primary endpoint.
The change in fibrosis risk scores | 3 months
  According to the Brunt criteria, fibrosis is classified in stages from stage 0 to stage 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt